CLINICAL TRIAL: NCT00801710
Title: CrossBoss and Stingray Catheter and Entera Guidewire Chronic Total Occlusion (CTO) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: BridgePoint Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-0001
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BridgePoint Medial System (Experimental)
  Interventions: Device: BridgePoint Medical System (CrossBoss Catheter, Stingray Catheter, Entera Guidewire)

INTERVENTIONS:
Device: BridgePoint Medical System (CrossBoss Catheter, Stingray Catheter, Entera Guidewire) — Revascularization of coronary artery chronic total occlusion.
  Use of the BridgePoint Medical System to cross coronary CTOs prior to definitive revascularization treatment via angioplasty and/or stent implant

SUMMARY:
This study is to determine if the BridgePoint Medical System (CrossBoss Catheter, Stingray Catheter, Entera Guidewire) can facilitate safe and effective placement of a guidewire in the true lumen of coronary vessels distal to a chronic total occlusion (CTO).

The hypothesis is that the BridgePoint Medical System can do this without an increase in major complications.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for coronary intervention
* de novo or restenotic CTO at least 3 months old, in proximal or mid coronary artery segment, 3.0-5.0 mm in diameter
* Mild/moderate proximal vessel tortuosity
* Mild/moderate lesion angulation
* Mild/moderate calcification
* Satisfactory distal vessel visualization
* Mild/moderate side branch interference
* 19 years old
* BMI<40
* LVEF>20%
* Signed informed consent

Exclusion Criteria:

* Extensive dissection from guidewire manipulation
* SVG or in-stent CTO
* Aorto-ostial CTO
* Unable to take aspirin, Clopidogrel, or Ticlopidine
* Thrombus/vessel filling defects
* Severe cerebrovascular disease/stroke within 1 month
* Intervention within 2 weeks
* Renal insufficiency
* GI bleeding
* Active infection
* Life expectancy <2 years
* Significant anemia
* Uncontrolled hypertension
* Severe electrolyte imbalance
* Anaphylaxis to contrast
* NYHA class IV
* Unstable angina requiring intervention
* MI within 2 weeks
* Uncontrolled diabetes
* Participating in another protocol
* Unwilling/unable to comply with protocol
* Angina/ischemia caused by target vessel

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
CTO Crossing Rate | Peri-procedural

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 30 days
Perforation rate | Peri-procedural
Acute myocardial infarction (AMI) | Peri-procedural

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — CardioVascular Center Frankfurt, St. Katharinen Hospital
Locations (4):
- Germany (4):
  - Main Taunus Hospital, Bad Soden
  - Klinikum Darmstadt, Darmstadt
  - CardioVascular Center Frankfurt, St. Katharinen Hospital, Frankfurt
  - Universitäres Herz- und Gefässzentrum Hamburg, Hamburg